CLINICAL TRIAL: NCT01211457
Title: A Phase I/II Combination Study of Sapacitabine in Acute Myeloid Leukemia or Myelodysplastic Syndromes
Brief Title: Study of Sapacitabine in Acute Myeloid Leukemia (AML) or Myelodysplastic Syndromes (MDS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYC682-11
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Sapacitabine; decitabine; venetoclax; elderly; AML; MDS; Refractory; relapsed; untreated
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence | interventions — sapacitabine; Decitabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sapacitabine/decitabine (Part 1 - completed) (Experimental): decitabine will be administered in alternating cycles with sapacitabine
  Interventions: Drug: sapacitabine and decitabine (Part 1 - completed)
- sapacitabine/venetoclax (Part 2 - recruiting) (Experimental): sapacitabine will be administered concomitantly with venetoclax
  Interventions: Drug: sapacitabine and venetoclax (Part 2 - recruiting)

INTERVENTIONS:
Drug: sapacitabine and decitabine (Part 1 - completed) — decitabine will be administered in alternating cycles with sapacitabine
  Arms: Sapacitabine/decitabine (Part 1 - completed)
Drug: sapacitabine and venetoclax (Part 2 - recruiting) — sapacitabine will be administered concomitantly with venetoclax
  Arms: sapacitabine/venetoclax (Part 2 - recruiting)

SUMMARY:
This is a combination study to evaluate sapacitabine administered in alternating cycles with decitabine in previously untreated Acute Myeloid Leukemia (AML) or concomitantly with venetoclax in previously treated AML or MDS

DETAILED DESCRIPTION:
This is an open-label, single arm, study of sapacitabine administered in alternating cycles with decitabine in elderly patients with previously untreated AML (Part 1) or concomitantly with venetoclax in adult patients with relapsed or refractory AML or MDS (Part 2). Treatment will be administered on an outpatient basis. One treatment cycle is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML based on WHO classification (Part 1) or previously treated AML or MDS (Part 2)
* Age 70 years or older for whom the treatment of choice is low-intensity therapy by investigator assessment or who has refused intensive induction therapy recommended by investigator (Part 1); age 18 years or older (Part 2)
* ECOG performance status 0-2
* Adequate renal function
* Adequate liver function
* Able to swallow capsules
* Ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* AML is of the sub-type of acute promyelocytic leukemia or extramedullary myeloid tumor without bone marrow involvement
* Known central nervous system (CNS) involvement by leukemia
* Uncontrolled intercurrent illness including
* Known hypersensitivity to decitabine (Part 1) or venetoclax (Part 2)
* Known to be HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2010-06-17 (Actual); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who achieve a clinical benefit response including CR, CRp, PR and major HI | 2 years

SECONDARY OUTCOMES:
response duration | 2 years
transfusion requirements | 2 years
hospitalized days | 2 years
overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M Kantarjian, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pooled Analysis of Elderly Patients with Newly Diagnosed AML Treated with Sapacitabine and Decitabine Administered in Alternating Cycles. Farhad Ravandi, Tapan M. Kadia, Gautam Borthakur, William G. Wierda, Stuart L. Goldberg, Meir Wetzler, Parameswaran Venugopal, Karen Seiter, Judy Chiao and Hagop M. Kantarjian. Blood 2012 120:2630.